CLINICAL TRIAL: NCT06363773
Title: Pilot, Exploratory, Prospective Study to Assess the Ability of Stereotactic Radiotherapy to Restore the Efficacy of Anti-PD1 Immunotherapy in Initially Long-responder Patients With Metastatic Progression.
Brief Title: A Study to Assess the Ability of Stereotactic Radiotherapy to Restore the Efficacy of Immunotherapy in Patients With Metastatic Cancer.
Acronym: RESTO-IMMUNO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESTO-IMMUNO; 2023-A02451-44 (Other: ANSM)
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Cancer
Keywords: stereotactic radiotherapy; immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Pilot, exploratory, prospective, monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic radiotherapy (Experimental): Patients will perform stereotactic radiotherapy with 3 sessions (8 Gy) during 20 minutes each and with 72 hours in-between, alongside anti-PD1 immunotherapy.
  Interventions: Radiation: Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy — Patients will perform stereotactic radiotherapy with 3 sessions (8 Gy) during 20 minutes each and with 72 hours in-between.
  Patients enrolled in the study would not have received this stereotactic radiotherapy outside the study, that is why this procedure is additional (compared to Standard of care) and considered as burdensome (as this is radiation). Before performing the stereotactic radiotherapy, patients will do a radiotherapy CT scanner (no injected) in order to prepare precisely the radiotherapy (treatment plan).

SUMMARY:
This study aims at enrolling patients with solid tumors at metastatic stage, considered long responders to immunotherapy (> 6 months) and displaying disease progression.

In this study, the investigator wants to evaluate specific modalities of stereotactic radiotherapy, with 3 sessions, each of 8 Gy, lasting 20 minutes and spaced 72 hours apart (Day 1, Day 4, Day 7). The radiotherapy device itself is not the subject of this study and will be used in accordance with its CE mark and indications.

The objective of the study is to assess the ability of stereotactic radiotherapy to restore the lost efficacy of immunotherapy. In particular, the abscopal effect will be assessed, i.e. the action of irradiating a particular target lesion and observing an effect on other distant metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older,
2. Patient with a metastatic solid tumor,
3. Patient with at least one target lesion (for radiotherapy) together with other secondary lesions that must be measurable,
4. Measurable disease according to RECIST 1.1 and iRECIST criteria,
5. Patient undergoing anti-PD1 immunotherapy as part of standard of care treatment,
6. Disease progression with immunotherapy (progression assessed by iRECIST criteria) but having received at least 6 months of immunotherapy,
7. Performance Status (PS) of 0 or 1,
8. Patient eligible for stereotactic radiotherapy,
9. Patient affiliated to or benefiting from a social security scheme,
10. Patient having been informed of the investigation and having signed the informed consent form prior to any study-specific procedures,
11. Patient willing and able to undergo all examinations and procedures in accordance with the clinical investigation plan.

Exclusion Criteria:

1. Patient having received previous radiotherapy since the start of immunotherapy,
2. Patient for whom first disease progression (pre-inclusion stage) is not confirmed secondarily (inclusion stage),
3. Patient with an active implantable medical device (e.g. pacemaker) or an active medical device worn on the body that could interact adversely with stereotactic radiotherapy treatment,
4. Patient with hematological cancer,
5. Symptomatic patient requiring a rapid change of systemic line according to the investigator's judgment,
6. Concurrent participation in another clinical trial, or patient having received an investigational product within 30 days prior to inclusion,
7. Pregnant or breast-feeding women,
8. Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate according to iRECIST criteria at 3 months after stereotactic radiotherapy in patients with confirmed progression after initial response to immunotherapy. | At 3 months after stereotactic radiotherapy
  Assessment of Objective Response Rate (Complete Response and Partial Response with iRECIST criteria) according to a centralised independent reading.

SECONDARY OUTCOMES:
Objective Response Rate according to RECIST 1.1 criteria at 3 months after stereotactic RT in patients with progression after initial response to immunotherapy. | At 3 months after stereotactic radiotherapy
  Assessment of Objective Response Rate (Complete Response and Partial Response with RECIST 1.1 criteria) according to a centralised independent reading.
Objective Response Rate according to iRECIST criteria up to 12 months after stereotactic radiotherapy in patients with confirmed progression after initial response to immunotherapy. | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to RECIST 1.1 criteria up to 12 months after stereotactic radiotherapy in patients with confirmed progression after initial response to immunotherapy. | Up to 12 months after stereotactic radiotherapy
Duration until new systemic treatment start. | Up to 12 months after stereotactic radiotherapy
  Duration (in days) before introduction of a new systemic treatment.
Incidence of Adverse Events (safety) | Up to 12 months after stereotactic radiotherapy
  Collection of adverse events (AEs) up to 12 months after radiotherapy.
Progression-Free Survival | Up to 12 months after stereotactic radiotherapy
Overall Survival | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to iRECIST criteria on the irradiated lesion only. | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to RECIST 1.1 criteria on the irradiated lesion only. | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to iRECIST criteria on all untreated lesion(s) (abscopal effect). | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to RECIST 1.1 criteria on all untreated lesion(s) (abscopal effect). | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to iRECIST criteria on each untreated lesion taken independently from others (abscopal effect). | Up to 12 months after stereotactic radiotherapy
Objective Response Rate according to RECIST 1.1 criteria on each untreated lesion taken independently from others (abscopal effect). | Up to 12 months after stereotactic radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Clinical, Soyaux, Charente, France

REFERENCES:
- [Result] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Result] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802
- [Result] Doyen J, Besse B, Texier M, Bonnet N, Levy A. PD-1 iNhibitor and chemotherapy with concurrent IRradiation at VAried tumor sites in advanced Non-small cell lung cAncer: the Prospective Randomized Phase 3 NIRVANA-Lung Trial. Clin Lung Cancer. 2022 May;23(3):e252-e256. doi: 10.1016/j.cllc.2021.10.008. Epub 2021 Oct 24. PMID 34810130
- [Result] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Result] Funck-Brentano E, Baghad B, Fort M, Aouidad I, Roger A, Beauchet A, Otmezguine Y, Blom A, Longvert C, Boru B, Saiag P. Efficacy of late concurrent hypofractionated radiotherapy in advanced melanoma patients failing anti-PD-1 monotherapy. Int J Cancer. 2020 Sep 15;147(6):1707-1714. doi: 10.1002/ijc.32934. Epub 2020 Feb 28. PMID 32083739
- [Result] Levy A, Khalifa J, Martin E, Botticella A, Quevrin C, Lavaud P, Aldea M, Besse B, Planchard D, Barlesi F, Deutsch E, Massabeau C, Doyen J, Le Pechoux C. Stereotactic body radiotherapy for extra-cranial oligoprogressive or oligorecurrent small-cell lung cancer. Clin Transl Radiat Oncol. 2023 May 3;41:100637. doi: 10.1016/j.ctro.2023.100637. eCollection 2023 Jul. PMID 37206411
- [Result] Ngwa W, Irabor OC, Schoenfeld JD, Hesser J, Demaria S, Formenti SC. Using immunotherapy to boost the abscopal effect. Nat Rev Cancer. 2018 May;18(5):313-322. doi: 10.1038/nrc.2018.6. Epub 2018 Feb 16. PMID 29449659
- [Result] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Result] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Result] Hatten SJ Jr, Lehrer EJ, Liao J, Sha CM, Trifiletti DM, Siva S, McBride SM, Palma D, Holder SL, Zaorsky NG. A Patient-Level Data Meta-analysis of the Abscopal Effect. Adv Radiat Oncol. 2022 Mar 3;7(3):100909. doi: 10.1016/j.adro.2022.100909. eCollection 2022 May-Jun. PMID 35372719
- [Result] Vanpouille-Box C, Alard A, Aryankalayil MJ, Sarfraz Y, Diamond JM, Schneider RJ, Inghirami G, Coleman CN, Formenti SC, Demaria S. DNA exonuclease Trex1 regulates radiotherapy-induced tumour immunogenicity. Nat Commun. 2017 Jun 9;8:15618. doi: 10.1038/ncomms15618. PMID 28598415
- [Result] Yasmin-Karim S, Ziberi B, Wirtz J, Bih N, Moreau M, Guthier R, Ainsworth V, Hesser J, Makrigiorgos GM, Chuong MD, Wei X, Nguyen PL, Ngwa W. Boosting the Abscopal Effect Using Immunogenic Biomaterials With Varying Radiation Therapy Field Sizes. Int J Radiat Oncol Biol Phys. 2022 Feb 1;112(2):475-486. doi: 10.1016/j.ijrobp.2021.09.010. Epub 2021 Sep 13. PMID 34530092